CLINICAL TRIAL: NCT01798589
Title: Clinical Evaluation of TRUE Test Ethylenediamine Dihydrochloride Allergen: Bioequivalence of Vehicle Formulations
Brief Title: Bioequivalence of Ethylenediamine Dihydrochloride Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allerderm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SPD 12 P1 401
Record Dates: First submitted 2013-02-20; First posted 2013-02-26 (Estimated); Results first posted 2020-05-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2020-05

CONDITIONS: Allergic Contact Dermatitis
Keywords: ethylenediamine dihydrochloride
MeSH Terms: conditions — Dermatitis, Allergic Contact

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ethylenediamine dihydrochloride (Experimental): Ethylenediamine dihydrochloride in methylcellulose 50 mcg/cm2 Ethylenediamine dihydrochloride in polyvinylpyrrolidone 50 mcg/cm2 Methylcellulose (negative control 1) Polyvinylpyrrolidone (negative control 2)
  Interventions: Drug: Ethylenediamine dihydrochloride allergen patch

INTERVENTIONS:
Drug: Ethylenediamine dihydrochloride allergen patch — 1 allergen panel containing 2 allergen and 2 control patches
  Other Names: T.R.U.E. Test allergen ethylenediamine dihydrochloride

SUMMARY:
The purpose of this study is to compare the allergen ethylenediamine dihydrochloride when prepared using methylcellulose versus preparation using polyvinylpyrrolidone.

DETAILED DESCRIPTION:
We propose an open, prospective, single-site study to evaluate the bioequivalence of ethylenediamine dihydrochloride in methylcellulose (MC)and polyvinylpyrrolidone (PVP) formulations. Bioequivalence will be determined in minimum of 15 adult subjects, with a clinical history of contact dermatitis and a positive patch test (current or previous) to ethylenediamine ("sensitives").

ELIGIBILITY:
Inclusion Criteria:

* Current or previous symptoms and/or history consistent with allergic contact dermatitis, and positive patch test (within the past 10 years) to ethylenediamine dihydrochloride
* 18 years of age or older, otherwise in good health
* Female subjects of childbearing potential must consent to a urine pregnancy test; results must be negative for study inclusion.
* Informed consent signed and understood by each subject.

Exclusion Criteria:

* Subjects unable to meet inclusion requirements
* Women who are breastfeeding or pregnant
* Topical treatment during the last 7 days with corticosteroids or other immunosuppressive agents on or near the test area
* Systemic treatment during the last 7 days with corticosteroids (equivalent to > 10 mg prednisone) or other immunosuppressive agents
* Treatment with ultraviolet (UV) light (including tanning) during the previous 3 weeks
* Acute dermatitis outbreak or dermatitis on or near the test area on the back
* Subjects unable to comply with patch test study requirements including multiple return visits and activity restrictions (e.g., protecting test panels from excess moisture due to showering or vigorous activity)
* Subject participation in clinical trials of investigational drugs, treatments, or devices, other than T.R.U.E. TEST, during this study or 3 weeks prior to inclusion in this study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Fowler, MD, Principal Investigator — Dermatology Specialists
Locations (1):
- Dermatology Specialists PSC, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects: All subjects were patched with 50 mcg/cm2 Ethylenediamine dihydrochloride in MC (methylcellulose), 50 mcg/cm2 Ethylenediamine dihydrochloride in PVP (polyvinylpyrrolidone) and negative controls
Period: Overall Study
Arm/Group | All Subjects
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Previous studies have indicated that enrollment of 15 subjects is sufficient to determine concordance and bioequivalence,
Groups:
- Ethylenediamine Dihydrochloride: Arm type: Experimental Ethylenediamine dihydrochloride in methylcellulose 50 mcg/cm2 Ethylenediamine dihydrochloride in polyvinylpyrrolidone 50 mcg/cm2 Methylcellulose (negative control 1) Polyvinylpyrrolidone (negative control 2)
  Ethylenediamine dihydrochloride: 1 allergen panel containing 2 allergen and 2 control patches
Arm/Group | Ethylenediamine Dihydrochloride
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16
Past Positive Response to Ethylenediamine [Number; unit: participants] | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Reactions to Ethylenediamine Dihydrochloride in MC (Methylcellulose) and Ethylenediamine Dihydrochloride in PVP (Polyvinylpyrrolidone)
Description: Bioequivalence will be calculated using concordance (Cohen's Kappa) between the number of subjects with positive reactions (defined as a score of 1+, 2+ or 3+) to 50 mcg/cm2 Ethylenediamine dihydrochloride in MC (methylcellulose) and 50 mcg/cm2 Ethylenediamine dihydrochloride in PVP (polyvinylpyrrolidone) and the number of subjects with negative reactions to 50 mcg/cm2 Ethylenediamine dihydrochloride in MC (methylcellulose) and 50 mcg/cm2 Ethylenediamine dihydrochloride in PVP (polyvinylpyrrolidone)
Time Frame: 21 days
Population: 16 subjects were enrolled. Data from 1 subject was not used in final analysis due to protocol deviation (out of window evaluation).
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects: Subjects were patched with a panel containing 50 mcg/cm2 Ethylenediamine dihydrochloride in MC (methylcellulose) vs 50 mcg/cm2 Ethylenediamine dihydrochloride in PVP (polyvinylpyrrolidone) and 2 negative controls
Arm/Group | All Subjects
Number analyzed (Participants) | 15
Participants
  Positive Reactions Ethylenediamine in MC | 10
  Positive Reactions Ethylenediamine in PVP | 11
Statistical Analysis 1: Comparison: All Subjects; Test type: Other — Bioequivalence is assessed based on concordance between the 2 allergen using Kappa statistic; Concordance = 66.7, 95% CI 2-sided [41.6 to 90.2]

2. Secondary Outcome: Number of Participants With Late Reactions to Ethylenediamine Dihydrochloride in MC (Methylcellulose) and Ethylenediamine Dihydrochloride in PVP (Polyvinylpyrrolidone)
Description: Number of subjects with a late reaction, defined as a positive reaction (score of 1+, 2+, 3+) initially appearing at 7-21 days after patch application)
Time Frame: Day 7-21
Population: Per protocol population
Measure: Number; unit: participants
Groups:
- All Subjects: All subjects were patched with a single panel containing ethylenediamine dihydrochloride, 50 mcg/cm2 in methylcellulose (MC), ethylenediamine dihydrochloride, 50 mcg/cm2 in polyvinlypyrrolidone (PVP) and 2 negative controls.
Arm/Group | All Subjects
Number analyzed (Participants) | 15
participants
  Late Reactions: Ethylenediamine in MC | 1
  Late Reactions Ethylenediamine in PVP | 1

3. Secondary Outcome: Number of Participants With Persistent Reactions to Ethylenediamine Dihydrochloride in MC (Methylcellulose) and Ethylenediamine Dihydrochloride in PVP (Polyvinylpyrrolidone)
Description: Number of subjects with a persistent reaction, defined as a positive reaction (score of 1+, 2+, 3+) initially appearing at one visit and persisting through the following visit.
Time Frame: Day 3-21
Population: Per protocol population
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 15
participants
  Persistent Reactions: Ethylenediamine in MC | 7
  Persistent Reactions Ethylenediamine in PVP | 8

4. Secondary Outcome: Number of Participants With Tape Irritation to Ethylenediamine Dihydrochloride in MC (Methylcellulose) and Ethylenediamine Dihydrochloride in PVP (Polyvinylpyrrolidone)
Description: Skin irritation associated with the adhesive tape (tape irritation) used to secure the test patches was evaluated at Visit 2 (day 2) 20 minutes following panel removal according to the following Tape Adhesion Score Scale: None (no irritation), Weak (faint to definite pink erythema), Moderate (moderate erythema, definite redness), Strong (severe erythema, very intense redness). Entire panel was scored as a whole- individual allergen sites were not scored separately.
Time Frame: Day 2 (48 hours after application)
Measure: Number; unit: participants
Groups:
- All Subjects: Tape Irritation, Day 2
Arm/Group | All Subjects
Number analyzed (Participants) | 15
participants
  No Tape Irritation | 10
  Weak Tape Irritation | 5
  Moderate Tape Irritation | 0
  Strong Tape Irritation | 0

5. Secondary Outcome: Number of Participants With Itching to Ethylenediamine Dihydrochloride in MC (Methylcellulose) and Ethylenediamine Dihydrochloride in PVP (Polyvinylpyrrolidone)
Description: Subject self-report of itching attributed to the test panels was recorded at Visit 2 (day 2), 20 minutes following panel removal. The following Itching Score Scale was used: None (no itching), Weak (minimal discomfort), Moderate (definite discomfort), Strong (significantly bothersome, possible interference with sleep or daily activity). Entire panel was scored as a whole- individual allergen sites were not scored separately.
Time Frame: Day 2 (48 hours after patch application)
Population: Per protocol
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects: Itching, Day 2
Arm/Group | All Subjects
Number analyzed (Participants) | 15
Participants
  No Itching | 6
  Weak Itching | 4
  Moderate Itching | 3
  Strong Itching | 2

6. Secondary Outcome: Number of Participants With Burning to Ethylenediamine Dihydrochloride in MC (Methylcellulose) and Ethylenediamine Dihydrochloride in PVP (Polyvinylpyrrolidone)
Description: Subject self-report of burning attributed to the test panels was recorded at Visit 2 (day 2), 20 minutes following panel removal. The following Burning Score scale was used: None (no burning), Weak (minimal discomfort), Moderate (definite discomfort), Strong (significantly bothersome, possible interference with sleep or daily activity). Entire panel was scored as a whole- individual allergen sites were not scored separately.
Time Frame: Day 2 (48 hours after application)
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Groups:
- Burning: Subject reported burning at day 2
Arm/Group | Burning
Number analyzed (Participants) | 15
Participants
  No Burning | 7
  Weak Burning | 6
  Moderate Burning | 1
  Strong Burning | 1

ADVERSE EVENTS:
Time Frame: Adverse Event information was collected for 21 days; from patch application at day 0 through the final visit at day 21. Two (2) adverse events (contact dermatitis and post-operative wound infection) were deemed by the Investigator, not related to use of the investigational allergens. The remaining adverse event, seborrhoeic dermatitis, could not be attributed to a single test allergen. Relationship in this case is to the allergen panel as a whole.
Groups:
- Ethylenediamine Hydrochloride: Adverse Events: Adverse events reported during clinical trial using investigational products: 50 mcg/cm2 Ethylenediamine dihydrochloride in MC (methylcellulose) and 50 mcg/cm2 Ethylenediamine dihydrochloride in PVP (polyvinylpyrrolidone)
Arm/Group | Ethylenediamine Hydrochloride: Adverse Events
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 3/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ethylenediamine Hydrochloride: Adverse Events (N=16)
Dermatitis, contact (Immune system disorders) | 1 (1)
Post operative wound infection (Infections and infestations) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No